CLINICAL TRIAL: NCT00597961
Title: Health Communication in Families
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 03-088
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer; Melanoma; Skin Cancer
Keywords: Lung; skin; melanoma
MeSH Terms: conditions — Lung Neoplasms; Melanoma; Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
There are two goals of this research study. First, we hope to develop a plan to guide family discussions that can help parents diagnosed with lung cancer talk about cancer risk with their adult children. Second, we want to understand how families talk about cancer prevention.

DETAILED DESCRIPTION:
In large part due to the advent of genetic testing, families have recently become a more central focus in cancer prevention. Given the high concordance of health behaviors within families (Kristeller et al., 1996), there is interest in developing family-wide behavior change interventions to reduce cancer risk. A cancer diagnosis represents a "teachable moment," in which a diagnosis may prompt health behavior change. Although this phenomenon has been observed among cancer survivors, it has not been examined among a patient's family members. Several critical questions exist about how families understand and communicate with regard to cancer risk information and what family processes facilitate or impede health behavior change. There is very little existent research in the area of cancer prevention among family members of cancer patients. Results in this area could help us develop interventions for family members who are motivated to make health behavior changes, and to inform and guide others who may not be motivated at the time their family member is diagnosed. Most importantly, the results could also help us intervene with family members of those who have been diagnosed with cancers where genetic and lifestyle components are important in the etiology of the illness, such as lung cancer and melanoma, and thus first-degree family members would benefit from strong messages to adopt healthy lifestyles. The research will rely on qualitative data collection and analysis. We will conduct qualitative interviews with 20 pairs of melanoma patients and one adult son or daughter, and 20 pairs of lung cancer patients and one adult child/sibling/or spouse. More specifically, for each pair of participants (i.e., the patient and his/her family member) we will conduct three interviews: an individual interview with the patient, an individual interview with the family member, and a joint interview where we will talk to the patient and family member at the same time. We will analyze interview data with a qualitative data computer analysis program, and identify themes and conclusions representing the core ideas in our data.

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer patients must have a history of smoking.
* Family members of lung cancer patients must be active smokers in order to participate in the study.
* All participants must be more than 18 years of age and be fluent in English.
* Patients must have received a diagnosis of either lung cancer or melanoma within the past 3 to 18 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Concentrating on two distinct tumor types, lung cancer and melanoma, because of the prominence of risk behaviors in the etiology of both of these cancers. With regard to lung cancer, we have identified high concordance of smoking among the spouses, siblings and children of recently diagnosed patients. In the context of melanoma, patients report a desire to use focused family discussions to encourage family members to reduce their skin cancer risk and increase early detection behaviors.
  "Family" defined as a group consisting of blood relatives, domestic partners, & on-blood relatives as defined by cancer patient. During interviews with melanoma-affected families we will be gathering data from a melanoma patient & ne of their adult sons or daughters. During the interviews with lung cancer-affected families we will be gathering data from a lung cancer patient and either one of their adult children, or one of their siblings, or their spouse.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2003-08-12 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
We will use data from our qualitative interviews to develop a family-focused assessment battery for examining risk perception and risk communication in families affected by cancer. | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ostroff, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org